CLINICAL TRIAL: NCT04851158
Title: Effectiveness of Two Different Methods on the Perceived Pain and Satisfaction During Intramuscular Antibiotic Injection: ShotBlocker and Local Vibration
Brief Title: Effectiveness of Two Different Methods During Intramuscular Antibiotic Injection: ShotBlocker, Local Vibration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Cemile Savcı, Assistant Professor, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20210067
Record Dates: First submitted 2021-03-19; First posted 2021-04-20 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Injections; Pain; Satisfaction, Patient
Keywords: Intramuscular injection; pain; ShotBlocker; local vibration; nursing
MeSH Terms: conditions — Pain; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: The sample size was determined as 35 persons for each group at the 0.5 effect size and 0.05 error level with the power analysis performed by taking into account the numerical values of the findings obtained from a previous study on this subject. ShotBlocker group:35; Local vibration group: 35; Control group:35 person
Who Masked: Participant
Masking Description: The sample of the study consisted of volunteer patients who applied to the adult emergency service, and who were administered antibiotics (amoxicillin / cefuroxime sodium) upon the physician's request, and who met the inclusion criteria of the study.
  Criteria for inclusion in the study:
  * Being over the age of 18,
  * Having no communication problem such as seeing, hearing and understanding problem,
  * Having no disease that can cause sensory loss,
  * Not having had IM injection in the last week,
  * Having no complication related to IM injections such as pain, abscess, infection, tissue necrosis, and hematoma at the injection site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ShotBlocker (Experimental): ShotBlocker will be used on 35 patients. For the patient group that is applied ShotBlocker, after cleansing the skin, the protruding surface of the device is placed facing the skin surface. The injection is applied with the appropriate technique, then ShotBlocker is removed and a light pressure is applied to the area with a cotton pad for 15-20 seconds.
  Interventions: Device: Effectiveness of ShotBlocker on the perceived pain and satisfaction during intramuscular antibiotic injection
- Local Vibration (Experimental): Local Vibration will be used on 35 patients. For the patient group that was subject to local vibration, local vibration was applied to the region with a vibrator for five minutes prior to injection, following a previous study on this subject. After that, 70% alcohol was used to cleanse the skin. The injection was applied with the appropriate technique, then a light pressure was applied to the area with a cotton pad for 15-20 seconds.
  Interventions: Device: Effectiveness of local vibrator device on the perceived pain and satisfaction during intramuscular antibiotic injection
- Control (No Intervention): For the control group (n=35), IM injection into the ventrogluteal region without using any tools is performed with the appropriate technique.

INTERVENTIONS:
Device: Effectiveness of ShotBlocker on the perceived pain and satisfaction during intramuscular antibiotic injection — Intervention: Verbal information was given to the participants prior to the intramuscular injection, and their written consents were obtained. The "Structured Information Form" consisting of five questions was applied by face-to-face interview method. Height and weight were measured, and BMI (kg/m2) was calculated and recorded in the "Structured Information Form".
  Application: ShotBlocker will be used on 35 patients during intramuscular injection.
  Final assessment: VAS will be applied immediately after the intramuscular injection to determine the pain and satisfaction levels of the participants.
  Arms: ShotBlocker
Device: Effectiveness of local vibrator device on the perceived pain and satisfaction during intramuscular antibiotic injection — Intervention: Verbal information was given to the participants prior to the intramuscular injection, and their written consents were obtained. The "Structured Information Form" consisting of five questions was applied by face-to-face interview method. Height and weight were measured, and BMI (kg/m2) was calculated and recorded in the "Structured Information Form".
  Application: Local vibrator device will be used on 35 patients during intramuscular injection.
  Final assessment: VAS will be applied immediately after the intramuscular injection to determine the pain and satisfaction levels of the participants.
  Arms: Local Vibration

SUMMARY:
In intramuscular injection applications, which are among the responsibilities and basic skills of nurses, different methods are used to reduce the pain caused by injection and increase the individual's satisfaction. ShotBlocker and local vibration are among the methods used for this purpose. The aim of the study is to examine the effectiveness of ShotBlocker and local vibration, which are among the non-pharmacological methods, on the perceived pain and satisfaction during ventrogluteal intramuscular antibiotic injection.

This randomized, controlled experimental study will be carried out in the adult emergency clinic of a training and research hospital in Istanbul between February and April 2021.

DETAILED DESCRIPTION:
The purpose of study was to evaluate four research hypotheses as follows:

H1: Using ShotBlocker during intramuscular antibiotic injection reduces the patient's injection pain.

H2: Using ShotBlocker during intramuscular antibiotic injection increases the patient's satisfaction with the injection.

H3: Using a local vibrator device during intramuscular antibiotic injection reduces the patient's injection pain.

H4: Using a local vibrator device during intramuscular antibiotic injection increases the patient's satisfaction with the injection.

Sampling of the Research: The sample number was determined at the 0.5 effect size and 0.05 error level with the power analysis performed by taking into account the numerical values of the findings obtained from a previous study on this subject. ShotBlocker group: 35; Local vibration group: 35, Control Group: 35 people.

The sample of the study will consist of volunteer patients who apply to the adult emergency department, who are administered antibiotics (amoxicillin / cefuroxime sodium) upon the physician's request, and who meet the inclusion criteria.

Data Collection Tools: Research data will be collected using the Structured Information Form created by the researchers, VAS Pain and VAS Satisfaction Scales.

Structured Information Form; Five questions regarding the descriptive characteristics of the participants (age, gender, body mass index (BMI), educational status, marital status) were included. BMI (kg/m2) of the participants will be calculated by the researcher.

Procedure:

1. Initial Assessment:

   Verbal information will be given to the participants and their written consents will be obtained prior to the intramuscular injection. The "Structured Information Form" consisting of five questions will be applied by face to face interview method, BMI will be calculated by measuring height and weight and recorded in the "Structured Information Form".

   ShotBlocker is a patented tool developed by Bionix (Toledo, OH, United States). It is a small, flat, horseshoe (U-shaped) shaped plastic tool with a thickness of 2 mm, which is used for pain control in intramuscular and subcutaneous injections, suitable for all age groups, has no known side effects, does not have drug properties, is non-invasive. Since it is not an invasive device, it is stated by the manufacturer that it can be used several times for the same patient after washing with soap. The protruding surface of the vehicle is placed in the area to be applied just before injection. Short blunt bumps on the surface of the vehicle do not pierce the skin.

   Local Vibrator one of the electric vibrator devices (dolphin massager device, 210-240 V, 50 Hz) produced by different brands was used. These devices with interchangeable heads have the ability to affect deep muscle groups, stimulate nerve endings and accelerate blood circulation thanks to mechanical vibration. During application, the device must be in full contact with the skin. Local vibration application reduces perceived pain by stimulating nerve fibers according to Melzack and Wall's Gate Control Theory.
2. Application:

   Before the drug is prepared, the physician's request will be checked by the researcher. Hands will be washed, the drug (amoxicillin / cefuroxime sodium) will be prepared by diluting with 4 ml of water for injection, the needle tip will be changed to 21G (0.8x40mm - green). The patient will be verbally informed, and the drug allergy status will be questioned. The patient will be asked to lie down in the prone position. The skin surface in the area where the IM injection will be applied will be observed by the researching specialist nurse for ecchymosis, scar, inflammation or edema. The presence of tenderness or stiffness will be evaluated by palpation, paying attention to muscle integrity. To the patient group who was applied local vibration; Before injection, local vibration will be applied to the region with a vibrator for five minutes, guided by a previous study on this subject. Afterwards, the skin will be cleaned using 70% alcohol and the injection will be applied with the appropriate technique, and then a light pressure will be applied to the area with a cotton pad for 15-20 seconds. For the patient group treated with ShotBlocker; After skin cleaning, the protruding surface of the vehicle will be placed facing the skin surface and the injection will be applied with the appropriate technique, then ShotBlocker will be removed and a light pressure will be applied to the area with a cotton pad for 15-20 seconds. In the control group; IM injection into the ventrogluteal area will be performed with the appropriate technique without using any tools.
3. Final Assessment:

The change from baseline in pain and satisfaction scores on the Visual Analogue Scale (VAS) will be measured immediately after intramuscular injection using VAS.

Ethical Considerations: The ethical compliance of the study was approved by the Istanbul Medeniyet University Goztepe Training and Research Hospital clinical research ethics committee (date and number: 10.02.2021/0067). Written institutional permission was obtained. After the purpose and duration of the study is explained, written informed consent is obtained from the patients on a voluntary basis.

Statistical Analyses: Data will be analyzed using SPSS (Statistical Package for Social Sciences, Chicago, Illinois) version 16.0.

Note: The research is not supported by any institution or organization.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 18, Having no communication problem such as seeing, hearing and understanding problem,
* Having no disease that can cause sensory loss,
* Not having had IM injection in the last week, Having no complication related to IM injections such as pain, abscess, infection, tissue necrosis, and hematoma at the injection site.

Exclusion Criteria:

Patients who do not meet the inclusion criteria will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Using ShotBlocker and local vibrator device during intramuscular antibiotic injection reduces the patient's injection related pain. | The procedure will take a total of 10 minutes.
  The change from baseline in pain scores will be measured immediately after intramuscular injection using Visual Analogue Scale (VAS) for pain. On a ten-centimetre long horizontal line, there are definitions of "no pain" at the left end and "unbearable pain" at the right end. High scores indicate a high level of pain.
Using ShotBlocker and local vibrator device during intramuscular antibiotic injection increases the patient's injection related satisfaction. | The procedure will take a total of 10 minutes.
  The change from baseline in satisfaction scores will be measured immediately after intramuscular injection using Visual Analogue Scale (VAS) for satisfaction. On a ten-centimetre long vertical line, there is the statement "Strongly dissatisfied" at the lower end of the line, and "Strongly satisfied" at the upper end. High scores indicate a high level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Kurtuluş Açıksarı, Study Chair — Göztepe Prof. Dr. Süleyman Yalçın City Hospital, Emergency Medicine Clinic; Alper Solakoğlu, Principal Investigator — Göztepe Prof. Dr. Süleyman Yalçın City Hospital, Emergency Medicine Clinic
Locations (1):
- Istanbul Medeniyet University Göztepe Prof. Dr. Süleyman Yalçın City Hospital, Emergency Medicine Clinic, Göztepe, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No